CLINICAL TRIAL: NCT00001169
Title: Clinical Investigation of Infections Due to Leishmanial Parasites
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 790144; 79-I-0144
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-02

CONDITIONS: Leishmaniasis; Leishmaniasis, Visceral
Keywords: Chemotherapy; Cytokines; Immunology; Kala-Azar; Leishmaniasis
MeSH Terms: conditions — Leishmaniasis; Leishmaniasis, Visceral

SUMMARY:
Mechanisms of host immune response to intracellular protozoa will be investigated in patients with naturally acquired infection employing a variety of in-vitro techniques. Both non-specific and antigen-specific humoral and cellular immune responses will be assessed. Parasites will be isolated from patients, cultivated in-vitro, and characterized. Responses to chemotherapy will be assessed parasitologically, immunologically and clinically.

DETAILED DESCRIPTION:
The main purpose of this protocol is to permit us to see patients who are referred to us for diagnosis and treatment of known or suspected leishmaniasis (from the Peace Corps, Smithsonian Institution, tourists, etc.). In the process of working up these patients, we sometimes encounter parasite isolates that are useful for research. We also can perform tests of cell-mediated immune function to evaluate how patients are responding to therapy. In addition, the protocol permits us to observe therapeutic responses to other drugs besides pentavalent antimony, if necessary.

ELIGIBILITY:
Must be between the ages of 1 and 65 years.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250
Dates: Start 1979-12; Study Completion 2001-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Ponce C, Ponce E, Morrison A, Cruz A, Kreutzer R, McMahon-Pratt D, Neva F. Leishmania donovani chagasi: new clinical variant of cutaneous leishmaniasis in Honduras. Lancet. 1991 Jan 12;337(8733):67-70. doi: 10.1016/0140-6736(91)90734-7. PMID 1670724
- [Background] Velasco O, Savarino SJ, Walton BC, Gam AA, Neva FA. Diffuse cutaneous leishmaniasis in Mexico. Am J Trop Med Hyg. 1989 Sep;41(3):280-8. PMID 2802018
- [Background] Badaro R, Falcoff E, Badaro FS, Carvalho EM, Pedral-Sampaio D, Barral A, Carvalho JS, Barral-Netto M, Brandely M, Silva L, et al. Treatment of visceral leishmaniasis with pentavalent antimony and interferon gamma. N Engl J Med. 1990 Jan 4;322(1):16-21. doi: 10.1056/NEJM199001043220104. PMID 2104665